CLINICAL TRIAL: NCT06451913
Title: Effect of Saccharomyces Boulardii CNCM I-745 on Gut Microbiota in Patients Undergoing Antibiotic Therapy (in the Context of Erythema Migrans (Early Skin Form of Lyme Borreliosis))
Acronym: SUBLYME
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Biocodex (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: SUBLYME - Sb 241; 2023-508694-80-01 (EU CTIS Number)
Record Dates: First submitted 2024-04-23; First posted 2024-06-11 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Erythema Migrans of Lyme Disease
Keywords: Erythema Migrans; Lyme Disease; Gut microbiota; Saccharomyces boulardii CNCM I-745; Lyme borreliosis
MeSH Terms: conditions — Erythema Chronicum Migrans; Glossitis, Benign Migratory; Lyme Disease | interventions — Amoxicillin

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, parallel-group, comparative study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The 2 types of investigational products will be checked for blind maintenance before release (capsules will be identical in size, shape, color and appearance). The principal investigator does not have access to the randomization (treatment) code, except in exceptional circumstances for valid medical or safety reason, such as occurrence of a serious adverse event for which the knowledge of the study medication would be considered essential for treating the patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Amoxicillin + Saccharomyces boulardii CNCM I-745 (Experimental): The patients will received oral Amoxicillin (1000 mg capsules bid) for 14 days and oral Saccharomyces boulardii CNCM I-745 (®) 250 mg x 2 capsules twice a day for 21 days.
  Interventions: Drug: Amoxicillin + Saccharomyces boulardii CNCM I-745; Other: Stool samples; Other: BSFS : Bristol Stool Form Scale; Other: GSRS : Gastrointestinal Symptom Rating Scale
- Amoxicillin + Placebo (Placebo Comparator): The patients will received oral Amoxicillin (1000 mg capsules bid) for 14 days + oral Placebo capsules for 21 days.
  Interventions: Drug: Amoxicillin + Placebo; Other: Stool samples; Other: BSFS : Bristol Stool Form Scale; Other: GSRS : Gastrointestinal Symptom Rating Scale

INTERVENTIONS:
Drug: Amoxicillin + Saccharomyces boulardii CNCM I-745 — At inclusion visit (V1), the Investigator will dispense and ask the subject to take Amoxicillin 1000 mg bid for 14 days + Saccharomyces boulardii 250 mg x 2 twice a day for 21 days
  Arms: Amoxicillin + Saccharomyces boulardii CNCM I-745
Drug: Amoxicillin + Placebo — At inclusion visit (V1),the Investigator will dispense and ask the subject to take Amoxicillin 1000 mg bid for 14 days + a matching placebo bid for 21 days
  Arms: Amoxicillin + Placebo
Other: Stool samples — The subject will be asked to collect thanks to four OMNIgene® •GUT OMR-200 kits :
  * an initial stool collection when returning home at D1 (in any case before any intake of amoxicillin and of the investigational medication and up to 1 day after D1).
  * a stool collection at home after the phone call 1, Day 7 (stool collection up to Day 7 + 1 day)
  * a stool collection at home after the phone call 2, Day 14 (stool collection up to Day 14 + 1 day)
  * at home the day of the Visit 2, Day 21 (stool collection up to Day 21 + 1 day)
Other: BSFS : Bristol Stool Form Scale — All included subjects will have to complete a stool diary BSFS (Bristol Stool Form Scale) daily and at each bowel movement, from Day 1 until the end of study treatment (Day 21). The patient will fill the form with the date, the time, and the stool texture.
Other: GSRS : Gastrointestinal Symptom Rating Scale — All included subjects will have to complete a GSRS (Gastrointestinal Symptom Response Score) questionnaire weekly from Day 1 until the end of the study treatment (Day 21).

SUMMARY:
The aim of this study is to assess the effect of Saccharomyces boulardii CNCM I-745 on gut microbiota in patients undergoing antibiotic therapy (in the context of erythema migrans (early skin form of Lyme borreliosis)).

DETAILED DESCRIPTION:
The study is designed to compare the efficacy of Saccharomyces boulardii CNCM-I-745 500 mg bid to a placebo in patients undergoing antibiotic therapy in the context of erythema migrans as the early form of Lyme borreliosis.

ELIGIBILITY:
Inclusion Criteria:

* Adult Patients, ≥18 years old.
* Who are prescribed antibiotic therapy (as per medical routine practices, amoxicillin 1000 mg bid for 14 days) in the context of erythema migrans (early skin form of Lyme borreliosis).
* Able to comply with study requirements and to provide signed informed consent before any study procedure.
* Has no condition that may interfere with the study assessments.
* Able to fulfil in the diary stool log, according to the physician's opinion.
* Regular defecation (frequency and stool consistency, with at least about three bowel movements a week).
* For women of childbearing potential:
* A negative urine pregnancy test immediately prior to starting the study treatment,
* Agreement to comply with approved methods of contraception during the whole study: unless they meet the criteria of post-menopausal, i.e. 12 months of spontaneous amenorrhea, women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, including women whose career, lifestyle, or sexual orientation precludes intercourse with a male partner, should use one or more acceptable methods of contraception that should be maintained throughout the study.

Exclusion Criteria:

* History of hypersensitivity to the study treatments (active substance or excipients), brewer's or baker's yeast,
* Contraindication and special warning to the study drugs according to the SmPCs,
* History of chronic constipation with passage of fewer than 3 spontaneous bowel movements per week on average,
* History of chronic or recurrent diarrhoea with spontaneous unformed bowel movements equivalent to or more often than 3 times daily,
* Prior gastrointestinal surgery (apart from appendectomy or cholecystectomy performed at least more than one year ago),
* History of Clostridium difficile infection,
* Active gastrointestinal inflammatory disease,
* Known chronic or recurrent systemic disorder that may interfere with the study drug evaluation,
* Immunocompromised (organtransplants, leukaemia, malignant tumours, radiotherapy, chemotherapy,prolonged high dose cortisone treatment, immunosuppressant treament) or critically ill patients (such as autoimmune disease, HIV,…), patients with a central venous catheter,
* Severe hepatic or renal impairment,
* Systemic antibacterial therapy during the 2 months prior to study enrollment,
* New prescription medications during the 2 weeks prior to study enrollment,
* Use of any drug or product that alters gut microbiota or function, such as probiotics, laxatives, antiemetics, cisapride, antisecretory or adsorbent treatments (racecadotril, smectite, activated charcoal), opiates such as loperamide, atropine and other cholinergic agents, 4 weeks prior to study enrollment and during the study,
* Intake of antifungals within 14 days prior to study enrollment,
* Substantial changes in eating habits within 30 days prior to receiving the first dose of IMP product, and during the study as assessed by the Investigator,
* History or presence of drug or alcohol abuse,
* Heavy smoker (more than 10 cigarettes per day),
* Breast-feeding woman,
* Patients enrolled in another interventional clinical trial where they received an investigation treatment within the past 30 days,
* Any condition or personal circumstance that, in the opinion of the investigator, rendered the subject unlikely or unable to comply with the full study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-07-16 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Assessment of the effect of Saccharomyces boulardii CNCM I-745, an antibiotic, and their combination on the gut microbiota of patients receiving antibiotic | At Day 1, Day 7, Day 14 and Day 21
  Primary endpoint : analysis of the intestinal microbiota in the patient's stools

SECONDARY OUTCOMES:
Assessment of the efficacy of Saccharomyces boulardii CNCM I-745 in prevention of antibiotic-associated diarrhoea (AAD) in patients undergoing antibiotic therapy | At Day 1, Day 7, Day 14 and Day 21
  Secondary efficacy endpoint : Incidence of AAD (The number of AAD episodes that occurred during the treatment period) will be assessed using the Bristol Stool Form Scale (BSFS) recorded daily.
Assessment of the efficacy of Saccharomyces boulardii CNCM I-745 on the stools in patients undergoing antibiotic therapy : Recorded stools in the Bristol Stool Form Scale (BSFS) | At Day 1, Day 7, Day 14 and Day 21
  Secondary efficacy endpoint : Time frame in hours up to the time of the last liquid or loose stool (defined as types 6 or 7 on Bristol Stool Form Scale (BSFS)) followed by the first 24-hour period with stool consistency improvement (no liquid or loose stool), as recorded by the patients in the stool diary or as collected by the investigator
Assess the effect of Saccharomyces boulardii CNCM I-745, an antibiotic, and their combination on the gastro-intestinal symptoms of patients receiving antibiotic therapy : Changes from baseline of the GSRS | Weekly from Day 1 to Day 21
  Secondary efficacy endpoint : Changes from baseline of the Gastrointestinal Symptom Rating Scale (GSRS) score (total score) and diarrhea sub-scores will be compared weekly between the treatment groups. The questionnaire, which contains 15 items, uses a seven-graded Likert scale, where 1 represents the most positive option and 7 the most negative one.

OTHER OUTCOMES:
Assessment of the safety and tolerability of Saccharomyces boulardii CNCM I-745. Recording adverse events | At each assessment time from baseline (Day 1 to Day 58)
  Safety endpoint : Recorded adverse events (number of events and number of participants with at least one event), vital signs, and physical examination
Assess the effect of Saccharomyces boulardii CNCM I-745, an antibiotic, and their combination on the specific gastro-intestinal symptoms of patients receiving antibiotic therapy : Gastrointestinal Symptom Rating scale (GSRS) | Weekly from Day 1 to Day 21
  Exploratory endpoint : Changes from baseline of the GSRS subscores (except diarrhea) will be compared weekly between the treatment groups.The questionnaire, which contains 15 items, uses a seven-graded Likert scale, where 1 represents the most positive option and 7 the most negative one.
Assess the effect of Saccharomyces boulardii CNCM I-745, an antibiotic, and their combination on the gut resistome of patients receiving antibiotic : Changes on the fecal Antimicrobial Resistance Genes (ARGs) | At Day 1, Day 7, Day 14 and Day 21
  Exploratory endpoint : Changes observed on the gut resistome, abundance and diversity of the fecal ARGs will be analysed by treatment group and at each assessment time.

CONTACTS AND LOCATIONS:
Overall Officials: Oana BERNARD, MD, Study Director — Chief Scientific Officer
Locations (1):
- University Medical Centre Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No